CLINICAL TRIAL: NCT00781001
Title: Efficacy of Inhaled Cannabis in Diabetic Painful Peripheral Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C06-SD-118
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Painful Diabetic Neuropathy
Keywords: neuropathic pain; diabetic neuropathy; cannabis; marijuana
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Placebo cannabis
  Interventions: Drug: Cannabis
- 2 (Experimental): Active cannabis - 1% THC by weight
  Interventions: Drug: Cannabis
- 3 (Experimental): Active cannabis - 4% THC by weight
  Interventions: Drug: Cannabis
- 4 (Experimental): Active cannabis - 7% THC by weight
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — 400mg placebo or active cannabis administered via the Volcano vaporizer 1x per study visit

SUMMARY:
The purpose of this study is to determine if vaporized cannabis is effective as an analgesic for the treatment of painful diabetic neuropathy.

DETAILED DESCRIPTION:
Neuropathic pain is caused by an insult to the nervous system and accounts for 25-50% of all pain clinic visits. Excluding low back pain, diabetic peripheral neuropathy is the most common neuropathic pain syndrome with an estimated prevalence of 600,000 cases in the United States. There are only 5 medications approved by the FDA for the treatment of neuropathic pain with only 2 out of the 5 approved for the treatment of diabetic peripheral neuropathy. Currently, there is a desperate need for more therapeutic agents for the treatment of neuropathic pain. We propose to use painful diabetic peripheral neuropathy (DPN) patients to study the efficacy of inhaled cannabis on neuropathic pain. We will enroll 20 subjects with each subject acting as their own control; receiving both placebo and three doses of inhaled aerosolized cannabis (low, medium, and high) in random order each separated by at least two weeks. Subjects will be assessed for reduction in pain, changes in normal sensation, changes in cognition, and effects of cannabis on experimentally induced pain.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* History of diabetes mellitus type 1 or type 2 who have stable glycemia and are maintained by diet or a stable regimen of diabetic therapy for at least 12 weeks prior to screening
* Painful diabetic peripheral neuropathy for at least 6 months prior to screening with symmetrical onset confirmed by neurological exam and a score of at least 3 on the investigator section (physical exam) of the MNSI (Michigan Neuropathy Screening Instrument) at screening.
* Subject has a pain rating of at least 4 on the 11 point Numeric Pain Scale.
* Patient is acceptable for enrollment as determined by the Investigator from the medical history, physical exam finding, 12 lead ECG findings, and clinical laboratory test results.
* HbA1C<11%.
* For female patients, a negative urine pregnancy test

Exclusion Criteria:

* Active opportunistic infections or opportunistic malignancies requiring acute treatment
* Current or past cannabis abuse/dependence, or current other psychoactive drug use disorder (e.g. opioids, methamphetamine, cocaine, alcohol)
* Presence of significant cardiac or pulmonary disease (e.g., tuberculosis, asthma)
* Pregnancy as ascertained by a self-report and a mandatory commercial pregnancy test before any marijuana or placebo consumption condition.
* Current serious mental illness--e.g. bipolar disorder, schizophrenia, or other psychotic disorder
* Other medical conditions that may lead to peripheral neuropathy
* Females who are pregnant or planning pregnancy.
* Females of child bearing potential not using a reliable means of birth control.
* Lower extremity amputations other than toes. Patients must not have phantom pain from amputated toes.
* Other painful conditions or pain of vascular origin that may confound the assessment of PDN.
* Subjects with unstable blood glucose level (Fasting< 70mg/dL or random blood glucose level > 250 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Spontaneous Pain Score | Baseline, 5, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 mins post-treatment

SECONDARY OUTCOMES:
Acute sensory threshold | Baseline, 5, 30, 60, 90, 120, 150, 180, 210, 240 mins post-treatment
Experimental pain score | Baseline, 5, 30, 60, 90, 120, 150, 180, 210, 240 mins post-treatment
Cognitive testing | Baseline, 60, 120, 240 mins post-treatment
Subjective highness | Baseline, 30, 60, 90, 120, 240 mins post-treatment
Adverse events | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Wallace, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, Hillcrest Medical Center, San Diego, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://www.cmcr.ucsd.edu